CLINICAL TRIAL: NCT03869190
Title: A Phase Ib/II, Open-Label, Multicenter, Randomized Umbrella Study Evaluating the Efficacy and Safety of Multiple Immunotherapy-Based Treatments and Combinations in Patients With Urothelial Carcinoma (MORPHEUS-UC)
Brief Title: Study Evaluating the Efficacy and Safety of Multiple Immunotherapy-Based Treatments and Combinations in Patients With Urothelial Carcinoma (MORPHEUS-UC)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Gilead Sciences, Inc., GlaxoSmithKline plc, Seattle Genetics and Astellas (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WO39613
Record Dates: First submitted 2019-03-08; First posted 2019-03-11 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Urothelial Carcinoma; Bladder Cancer
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms | interventions — atezolizumab; enfortumab vedotin; niraparib; magrolimab; Tiragolumab; sacituzumab govitecan; tocilizumab; Cisplatin; Gemcitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (16):
- Atezolizumab for mUC Cohort (Stage 1) (Active Comparator): Participants will receive atezolizumab until unacceptable toxicity or loss of clinical benefit, as determined by the investigator after an integrated assessment of radiographic and biochemical data, local biopsy results (if available), and clinical status.
  Enrollment is closed.
  Interventions: Drug: Atezolizumab
- Atezolizumab + Enfortumab Vedotin for mUC Cohort (Stage 1) (Experimental): Participants will receive atezolizumab and Enfortumab Vedotin (EV) until unacceptable toxicity or loss of clinical benefit, as determined by the investigator after an integrated assessment of radiographic and biochemical data, local biopsy results (if available), and clinical status. Enrollment is closed.
  Interventions: Drug: Atezolizumab; Drug: Enfortumab Vedotin
- Atezolizumab + Niraparib for mUC Cohort (Stage 1) (Experimental): Participants will receive atezolizumab and Niraparib (Nira) until unacceptable toxicity or loss of clinical benefit, as determined by the investigator after an integrated assessment of radiographic and biochemical data, local biopsy results (if available), and clinical status. Enrollment is closed.
  Interventions: Drug: Atezolizumab; Drug: Niraparib
- Atezolizumab + Magrolimab for mUC Cohort (Stage 1) (Experimental): Participants will receive atezolizumab and magrolimab (Hu5F9-G4) until unacceptable toxicity or loss of clinical benefit, as determined by the investigator after an integrated assessment of radiographic and biochemical data, local biopsy results (if available), and clinical status. Enrollment is closed.
  Interventions: Drug: Atezolizumab; Drug: Magrolimab (Hu5F9-G4)
- Atezolizumab + Tiragolumab for mUC Cohort (Stage 1) (Experimental): Participants will receive atezolizumab and Tiragolumab (Tira) until unacceptable toxicity or loss of clinical benefit, as determined by the investigator after an integrated assessment of radiographic and biochemical data, local biopsy results (if available), and clinical status. Enrollment is closed.
  Interventions: Drug: Atezolizumab; Drug: Tiragolumab
- Atezolizumab + Sacituzumab Govitecan for mUC Cohort (Stage 1) (Experimental): Participants will receive atezolizumab and Sacituzumab Govitecan (SG) until unacceptable toxicity or loss of clinical benefit, as determined by the investigator after an integrated assessment of radiographic and biochemical data, local biopsy results (if available), and clinical status. Enrollment is closed.
  Interventions: Drug: Atezolizumab; Drug: Sacituzumab Govitecan
- Atezolizumab + Tocilizumab for mUC Cohort (Stage 1) (Experimental): Participants will receive atezolizumab and Tocilizumab (TCZ) until unacceptable toxicity or loss of clinical benefit, as determined by the investigator after an integrated assessment of radiographic and biochemical data, local biopsy results (if available), and clinical status. Enrollment is closed.
  Interventions: Drug: Atezolizumab; Drug: Tocilizumab
- Atezolizumab + RO7122290 for mUC Cohort (Stage 1) (Experimental): Participants will receive atezolizumab and RO7122290 until unacceptable toxicity or loss of clinical benefit, as determined by the investigator after an integrated assessment of radiographic and biochemical data, local biopsy results (if available), and clinical status. Enrollment is closed.
  Interventions: Drug: Atezolizumab
- Atezolizumab + Enfortumab Vedotin for mUC Cohort (Stage 2) (Experimental): Participants will receive atezolizumab and Enfortumab Vedotin (EV) until unacceptable toxicity or loss of clinical benefit, as determined by the investigator after an integrated assessment of radiographic and biochemical data, local biopsy results (if available), and clinical status. Enrollment is closed.
  Interventions: Drug: Atezolizumab; Drug: Enfortumab Vedotin
- Atezolizumab + Sacituzumab Govitecan for mUC Cohort (Stage 2) (Experimental): Participants will receive atezolizumab and Sacituzumab Govitecan (SG) until unacceptable toxicity or loss of clinical benefit, as determined by the investigator after an integrated assessment of radiographic and biochemical data, local biopsy results (if available), and clinical status. Enrollment is closed.
  Interventions: Drug: Atezolizumab; Drug: Sacituzumab Govitecan
- Atezolizumab for Cisplatin-ineligible MIBC Cohort 1 PD-L1+ Arm 1 (Active Comparator): Participants will receive Atezolizumab for 3 cycles pre-surgery and 14 cycles post-surgery.
  Interventions: Drug: Atezolizumab
- Atezolizumab + Tiragolumab for Cisplatin-ineligible MIBC Cohort 1 PD-L1+ Arm 2 (Experimental): Participants will receive Atezolizumab and Tiragolumab (Tira) for 3 cycles pre-surgery and 14 cycles post-surgery.
  Interventions: Drug: Atezolizumab; Drug: Tiragolumab
- Atezolizumab for Cisplatin-ineligible MIBC Cohort 2 PD-L1- Arm 1 (Active Comparator): Participants will receive Atezolizumab for 3 cycles pre-surgery and 14 cycles post-surgery.
  Interventions: Drug: Atezolizumab
- Atezolizumab + Tiragolumab for Cisplatin-ineligible MIBC Cohort 2 PD-L1- Arm 2 (Experimental): Participants will receive Atezolizumab and Tiragolumab (Tira) for 3 cycles pre-surgery and 14 cycles post-surgery.
  Interventions: Drug: Atezolizumab; Drug: Tiragolumab
- Cisplatin-eligible MIBC Cohort 3 Arm 1 (Active Comparator): Participants will receive 3 cycles of Atezolizumab, Cisplatin, and Gemcitabine pre-surgery and 14 cycles of Atezolizumab only post-surgery.
  Interventions: Drug: Atezolizumab; Drug: Cisplatin; Drug: Gemcitabine
- Cisplatin-eligible MIBC Cohort 3 Arm 2 (Experimental): Participants will receive Atezolizumab, Tiragolumab (Tira), Cisplatin and Gemcitabine for 3 cycles pre-surgery and 14 cycles of Atezolizumab and Tiragolumab (Tira) post-surgery.
  Interventions: Drug: Atezolizumab; Drug: Tiragolumab; Drug: Cisplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: Atezolizumab — For the control, + EV, + Nira, + Tira, and + SG arms, + RO7122290, Atezolizumab will be administered intravenously (IV) at a fixed dose of 1200 mg every 3 weeks (Q3W) on Day 1 of each 21-day cycle.
  For the Atezo + Hu5F9-G4 and + TCZ arms, Atezo will be administered IV at a fixed dose of 840 mg every 2 weeks (Q2W) on Days 1 and 15 of each 28-day cycle.
Drug: Enfortumab Vedotin — Enfortumab vedotin will be administered at a dose of 1.25 mg/kg IV on Days 1 and 8 of each 21-day cycle.
  Arms: Atezolizumab + Enfortumab Vedotin for mUC Cohort (Stage 1); Atezolizumab + Enfortumab Vedotin for mUC Cohort (Stage 2)
Drug: Niraparib — Niraparib will be administered at a dose of 200 mg once daily (QD) by mouth.
  Arms: Atezolizumab + Niraparib for mUC Cohort (Stage 1)
Drug: Magrolimab (Hu5F9-G4) — Participants will receive an 1-mg/kg priming dose IV on Day 1 followed by three weekly IV doses of 30 mg/kg on Days 8, 15, and 22. During Cycle 2, participants will receive weekly IV doses of 30 mg/kg on Days 1, 8, 15, and 22. For all subsequent cycles, participants will receive 30 mg/kg on Days 1 and 15. Cycle = 28 days.
  Arms: Atezolizumab + Magrolimab for mUC Cohort (Stage 1)
Drug: Tiragolumab — Tiragolumab will be administered at a dose of 600 mg IV on Day 1 of each 21-day cycle.
  Arms: Atezolizumab + Tiragolumab for Cisplatin-ineligible MIBC Cohort 1 PD-L1+ Arm 2; Atezolizumab + Tiragolumab for Cisplatin-ineligible MIBC Cohort 2 PD-L1- Arm 2; Atezolizumab + Tiragolumab for mUC Cohort (Stage 1); Cisplatin-eligible MIBC Cohort 3 Arm 2
Drug: Sacituzumab Govitecan — Sacituzumab Govitecan will be administered at a dose of 10 mg/kg by IV on Day 1 and 8 of each 21-day cycle.
  Arms: Atezolizumab + Sacituzumab Govitecan for mUC Cohort (Stage 1); Atezolizumab + Sacituzumab Govitecan for mUC Cohort (Stage 2)
Drug: Tocilizumab — Tocilizumab will be administered by IV infusion at a dose of 8 mg/kg every 4 weeks (Q4W) on Day 1 of each 28-day cycle.
  Arms: Atezolizumab + Tocilizumab for mUC Cohort (Stage 1)
Drug: Cisplatin — Cisplatin will be administered at a dose of 70mg/m^2 by IV on Day 1 of each cycle for Cycles 1-3 pre-surgery.
  Arms: Cisplatin-eligible MIBC Cohort 3 Arm 1; Cisplatin-eligible MIBC Cohort 3 Arm 2
Drug: Gemcitabine — Gemcitabine will be administered at a dose of 1000mg/m^2 by IV on Days 1 and 8 of each cycle for Cycles 1-3 pre-surgery.
  Arms: Cisplatin-eligible MIBC Cohort 3 Arm 1; Cisplatin-eligible MIBC Cohort 3 Arm 2

SUMMARY:
A Phase Ib/II, open-label, multicenter, randomized, umbrella study in participants with MIBC and in participants with locally advanced or metastatic Urothelial Carcinoma (UC) who have progressed during or following a platinum-containing regimen. The study is designed with the flexibility to open new treatment arms as new treatments become available, close existing treatment arms that demonstrate minimal clinical activity or unacceptable toxicity, or modify the participant population (e.g., with regard to prior anti-cancer treatment or biomarker status). Participants in the mUC Cohort who experience loss of clinical benefit or unacceptable toxicity during Stage 1 may be eligible to continue treatment with a different treatment regimen for Stage 2.

ELIGIBILITY:
Inclusion Criteria for mUC Cohort:

* Histologically documented, locally advanced or metastatic UC (also termed TCC or urothelial cell carcinoma of the urinary tract; including renal pelvis, ureters, urinary bladder, and urethra)
* Availability of a representative tumor specimen that is suitable for determination of PD-L1 and/or additional biomarker status by means of central testing
* Disease progression during or following treatment with no more than one platinum-containing regimen for inoperable, locally advanced or metastatic UC or disease recurrence
* ECOG Performance Status of 0 or 1
* Measurable disease (at least one target lesion) according to RECIST v1.1
* Adequate hematologic and end-organ function
* Negative HIV test at screening
* Negative total hepatitis B core antibody (HBcAb) test and hepatitis C virus (HCV) antibody at screening
* Tumor accessible for biopsy
* For women of childbearing potential: agreement to remain abstinent or use contraceptive measures and agreement to refrain from donating eggs
* For men: agreement to remain abstinent or use contraceptive measures, and agreement to refrain from donating sperm

Inclusion Criteria for MIBC Cohorts:

* ECOG PS of 0 or 1
* Fit and planned-for cystectomy
* Histologically documented MIBC (pT2-4, N0, M0), also termed TCC or urothelial cell carcinoma of the urinary bladder
* N0 or M0 disease by CT or MRI
* Adequate hematologic and end-organ function
* Availability of TURBT specimen
* Negative HIV, HBcAb, and HCV test at screening
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures and agreement to refrain from donating eggs as outlined for each specific treatment arm
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm, as outlined for each specific treatment arm

Exclusion Criteria for mUC Cohort:

* Prior treatment with a T-cell co-stimulating therapy or a CPI including anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies
* Prior treatment with any of the protocol-specified study treatments including treatment with poly (adenosine diphosphate [ADP]-ribose) polymerase (PARP) inhibitor, nectin-4 targeting agents, signal regulatory protein alpha-targeting agents, or TIGIT-targeting agents, Trop-2 targeting agents, FAP-directed therapies, 4-1BB (CD137)-directed therapies, or topoisomerase 1 inhibitors
* Treatment with investigational therapy within 28 days prior to initiation of study treatment
* Any approved anti-cancer therapy, including chemotherapy or hormonal therapy, within 3 weeks prior to initiation of study treatment
* Eligibility only for the control arm
* Prior allogeneic stem cell or solid organ transplantation
* Treatment with systemic immunostimulatory agents within 4 weeks or 5 half-lives of the drug (whichever is longer) prior to the initiation of study treatment
* Treatment with systemic immunosuppressive medication within 2 weeks prior to initiation of study treatment or anticipation of need for systemic immunosuppressant medication during study treatment
* Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during atezolizumab treatment or within 5 months after the last dose of atezolizumab
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures
* Uncontrolled tumor-related pain
* Uncontrolled or symptomatic hypercalcemia
* Symptomatic, untreated, or actively progressing CNS metastases
* History of leptomeningeal disease
* Active or history of autoimmune disease or immune deficiency
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis
* History of malignancy other than UC within 2 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death
* Active tuberculosis
* Severe infection within 4 weeks prior to initiation of study treatment
* Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment
* Significant cardiovascular disease
* Uncontrolled hypertension
* Grade 3 or greater hemorrhage or bleeding event within 28 days prior to initiation of study treatment
* Major surgical procedure, other than for diagnosis, within 4 weeks prior to initiation of study treatment
* Pregnancy or breastfeeding, or intention of becoming pregnant during the study
* Additional drug-specific exclusion criteria might apply

Exclusion for MIBC Cohorts:

* Prior treatment with systemic immunostimulatory agents prior to the initiation of study treatment
* Eligibility only for the control arm
* Prior allogeneic stem cell or solid organ transplantation
* Treatment with systemic immunosuppressive medication within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressant medication during study treatment, with the following exceptions: Patients who received acute, low-dose, systemic immunosuppressant medications, or a one-time pulse dose of systemic immunosuppressant medication are eligible for the study after Medical Monitor approval has been obtained. Patients who received mineralocorticoids, corticosteroids for chronic obstructive pulmonary disease or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study.
* Severe infection within 4 weeks prior to initiation of study treatment
* Pregnancy or breastfeeding, or intention of becoming pregnant during the study
* Also includes all the mUC exclusion criteria

Additional Exclusion Criteria for Atezo+Tira and Atezo (Atezolizumab) +Tira+Cis (Cisplatin)+Gem (Gemcitabine) in the MIBC Cohorts:

- Active Epstein-Barr virus (EBV) infection or known or suspected chronic active EBV infection at screening.

Additional Exclusion Criteria for the Cisplatin-Eligible MIBC Cohort:

* Patients who decline neoadjuvant cisplatin-based chemotherapy or in whom neoadjuvant cisplatin-based therapy is not appropriate.
* Impaired renal function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2025-10-08 (Actual); Study Completion 2025-12-22 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) for mUC Cohort Stage 1 | Baseline until disease progression or loss of clinical benefit (approximately 5-7 years)
  Objective response rate, defined as the proportion of participants with a CR or PR on two consecutive occasions >=4 weeks apart during Stage 1, as determined by the investigator according to RECIST v1.1.
pCR for Muscle Invasive Bladder Cancer (MIBC) Cohorts | Randomization to approximately 5-7 years
  pCR, defined as the proportion of participants with an absence of residual invasive cancer of the complete resected specimen.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) for mUC Cohort Stage 1 | Randomization until the first occurrence of disease progression or death from any cause, which ever occurs first, through the end of study (approximately 5-7 years) as determined by the investigator according to RECIST 1.1
  PFS after randomization, defined as the time from randomization to the first occurrence of disease progression or death from any cause (whichever occurs first) in Stage 1, as determined by the investigator according to RECIST v1.1.
Overall Survival (OS) for mUC Cohort Stage 1 | Randomization to death from any cause, through the end of study (approximately 5-7 years)
  OS after randomization,defined as the time from randomization to death from any cause.
Overall Survival (at specific time-points) for mUC Cohort Stage 1 | 12 months
  OS rate at specific timepoints, defined as the proportion of patients who have not experienced death from any cause at that timepoint.
Duration of Response (DOR) for mUC Cohort Stage 1 | Randomization until first occurrence of a documented objective response to the first recorded occurrence of disease progression or death from any cause (whichever occurs first), through end of study (approximately 5-7 years)
  DOR, defined as the time from the first occurrence of a documented objective response during Stage 1 to disease progression or death from anycause (whichever occurs first), as determined by the investigator according to RECIST v1.1.
Disease Control Rate (DCR) for mUC Cohort Stage 1 | Baseline through end of study (approximately 5-7 years)
  Disease control, defined as stable disease >= 18 weeks or a CR or PR, as determined by the investigator according to RECIST v1.1.
Percentage of Participants with Adverse Events for mUC Cohort Stage 1 | Baseline to end of study (approximately 5-7 years)
Serum Concentration of Atezolizumab for mUC Cohort Stage 2 | At pre-defined intervals from first administration of study drug up to approximately 5-7 years
Serum Concentration of Enfortumab Vedotin for mUC Cohort Stage 2 | At pre-defined intervals from first administration of study drug up to approximately 5-7 years
Serum Concentration of Sacituzumab Govitecan for mUC Cohort Stage 2 | At pre-defined intervals from first administration of study drug up to approximately 5-7 years
Presence of ADAs to Atezolizumab for mUC Cohort Stage 2 | Baseline to approximately 5-7 years
  For drugs for which ADA formation is measured: presence of ADAs during the study relative to the presence of ADAs at baseline.
Percentage of Participants with Adverse Events for mUC Cohort Stage 2 | Baseline to end of study (approximately 5-7 years)
Landmark Recurrence-Free Survival (RFS) for MIBC Cohorts | 12, 18, 24 months
  Landmark RFS, defined as RFS at specific timepoints.
Landmark Event-Free Survival (EFS) for MIBC Cohorts | 12, 18, 24 months
  Landmark EFS, defined as EFS at specific timepoints.
Landmark Overall Survival (OS) for MIBC Cohorts | 12, 18, 24 months
  Landmark OS, defined as OS at specific timepoints.
Percentage of Participants with Adverse Events for MIBC Cohorts | Baseline to approximately 5-7 years

CONTACTS AND LOCATIONS:
Locations (33):
- United States (10):
  - UCLA Department of Medicine, Los Angeles, California
  - UCSF Comprehensive Cancer Ctr, San Francisco, California
  - Stanford Cancer Center, Stanford, California
  - University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Norton Cancer Institute, Louisville, Kentucky
  - Memorial Sloan-Kettering Cancer Center, Commack, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- France (4):
  - Centre Francois Baclesse, Caen
  - Centre Leon Berard, Lyon
  - Institut régional du Cancer Montpellier, Montpellier
  - Institut Claudius Regaud, Toulouse
- Greece (2):
  - Attiko Hospital University of Athens, Athens
  - Athens Medical Center, Athens
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Severance Hospital, Seoul
- Spain (12):
  - Complejo Hospitalario Universitario de Santiago (CHUS), Santiago de Compostela, LA Coruna
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - Vall d?Hebron Institute of Oncology (VHIO), Barcelona, Barcelona
  - Hospital Clinic i Provincial, Barcelona
  - Institut Catala d Oncologia Hospitalet, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital General Universitario Gregorio Mara, Madrid
  - MD Anderson Cancer Center, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz., Madrid
  - Hospital Univ 12 de Octubre, Madrid
  - START Madrid. Centro Integral Oncologico Clara Campal, Madrid
  - Hospital Clinico Universitario de Valencia, Valencia
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan
- Royal Marsden NHS Foundation Trust, Sutton, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Drakaki A, Powles T, Bamias A, Martin-Liberal J, Shin SJ, Friedlander T, Tosi D, Park C, Gomez-Roca C, Joly Lobbedez F, Castellano D, Morales-Barrera R, Moreno-Candilejo I, Flechon A, Yuen K, Rishipathak D, DuPree K, Young F, Michielin F, Shemesh CS, Steinberg EE, Williams P, Lee JL. Atezolizumab plus Magrolimab, Niraparib, or Tocilizumab versus Atezolizumab Monotherapy in Platinum-Refractory Metastatic Urothelial Carcinoma: A Phase Ib/II Open-Label, Multicenter, Randomized Umbrella Study (MORPHEUS Urothelial Carcinoma). Clin Cancer Res. 2023 Nov 1;29(21):4373-4384. doi: 10.1158/1078-0432.CCR-23-0798. PMID 37651261